CLINICAL TRIAL: NCT04158089
Title: Holistic Assessment of Tulsa Children's Health
Acronym: HATCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: Oklahoma Center for the Advancement of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: HS1871
Record Dates: First submitted 2019-10-29; First posted 2019-11-08 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Pregnancy

STUDY DESIGN:
Intervention Model Description: This intervention examines whether the use of texted attachment exercises to effectively increase maternal prenatal bonding.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Due to the behavioral design of the intervention, it is impossible to mask participants (who are asked to do tasks) or investigators (who train participants and contact them about tasks). However, care providers are not involved in the study, and the statistical analyses will be conducted with a de-identified data set.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No intervention (No Intervention): Participants in the "No intervention" group will receive treatment (e.g., prenatal care) as usual.
- Attachment Exercises (Experimental): Participants in the "Attachment Exercises" group will receive daily texts over the 2-week intervention period with activities to do from home that are designed to increase feelings of attachment (e.g., read a children's book aloud; sing a nursery rhyme; picture giving the baby a bath; tell the baby a story; etc.).
  Interventions: Behavioral: Babies and Moms connected through Love, Openness, and Opportunity (BLOOM)

INTERVENTIONS:
Behavioral: Babies and Moms connected through Love, Openness, and Opportunity (BLOOM) — Participants will be randomly assigned into one of two groups for the BLOOM intervention; the control group will receive treatment as usual. Participants assigned to the treatment group will receive texted attachment exercises to complete from home. The intervention will take place over a 2-week period. Participants in the "Attachment Exercises" group will receive a text every day with an activity designed to increase feelings of attachment (e.g., read a children's book; sign a nursery rhyme; picture giving your baby a baby; tell your baby a story, etc.).
  Arms: Attachment Exercises

SUMMARY:
The primary goal of this study is to rapidly increase maternal-fetal bonding, a strong predictor of maternal health practices during pregnancy, through an intervention, BLOOM (Babies and Moms, connected by Love, Openness, and Opportunity). Specifically, the investigators will examine change in maternal-fetal bonding across pregnancy and implications for change in maternal smoking during pregnancy using a randomized clinical trial design in a longitudinal, multi-ethnic cohort study of 160 women (ages 18 or older) who are 12-16 weeks pregnant. Participants will be randomly assigned into one of two groups for the intervention; the control group will receive treatment as usual. Participants assigned to the treatment group will receive texted attachment/mindfulness exercises. Participants will complete an in-depth initial assessment that includes sociodemographic measures as well as a battery to capture maternal-fetal bonding and self-reported smoking. Pre- and post-tests will be used to assess maternal-fetal bonding and smoking before and after the intervention to allow for examination of change across pregnancy. The positive impacts of this work include information that will be used to reduce the impact of unintended pregnancy for adverse infant health outcomes.

DETAILED DESCRIPTION:
Unintended pregnancy (unwanted and/or mistimed pregnancy) heightens the risk for adverse birth outcomes, including preterm birth and very low birth weight (< 1500 grams), which have significant public health costs. Despite decades spent attempting to reduce the proportion of pregnancies that are unintended, nearly half (45%) of all pregnancies are unintended. Among women living in poverty, rates of unintended pregnancy are considerably higher. In this study, investigators focus instead on the reduction of a risky maternal health practice associated with adverse birth outcomes that are more common when pregnancies are unintended: maternal prenatal smoking. The study focuses on rapidly increasing maternal-fetal bonding, a mediator of the relationship between unintended pregnancy and maternal health practices during pregnancy, through a recently piloted intervention, BLOOM (Babies and Moms, connected by Love, Openness, and Opportunity). Specifically, the investigators will examine change in maternal-fetal bonding across pregnancy and implications for change in maternal smoking during pregnancy. The proposed study will use a randomized clinical trial design in a longitudinal, multi-ethnic cohort study of 160 predominately low-income women (ages 18 or older) who are 12-16 weeks pregnant and planning to continue their pregnancies and be primary caregivers to their infants. Participants will be randomly assigned into one of two groups for the intervention; the control group will receive treatment as usual. Participants assigned to the treatment group will receive texted attachment/mindfulness exercises. Participants will complete an in-depth initial assessment that includes sociodemographic measures as well as a battery to capture maternal-fetal bonding and self-reported smoking. The 2-week intervention will be conducted within two weeks following Assessment 1. Participants will then be asked to complete a follow-up survey near the beginning of their 3rd trimester to assess maternal-fetal bonding and smoking to allow for examination of change across pregnancy. Impacts of prior interventions to reduce unintended pregnancy and its associated adverse infant outcomes have been modest; reducing the negative association between unintended pregnancy and adverse outcomes through enhancing maternal prenatal attachment makes this project highly significant. This project will be the first to target maternal-fetal bonding through the use of a cellphone-based intervention designed to increase feelings of bonding through attachment and mindfulness exercises, making it highly innovative. The positive impacts of this work include information that will be used to reduce the impact of unintended pregnancy for adverse infant health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Between 12-16 weeks pregnant at the time of enrollment.

Exclusion Criteria:

* Unable to communicate in either English or Spanish
* Planning to either terminate the pregnancy or place the baby for adoption.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2021-12-20 (Actual); Primary Completion 2023-07-18 (Actual); Study Completion 2023-07-18 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Maternal-Fetal Attachment at 4 months | Through study completion, an average of 1 year
  Maternal-Fetal Attachment Scale (MFAS) is a 24-item, Likert type, self-rated scale with five subscales (Cranley, 1981)
Change from Baseline Self-Reported Smoking Status at 4 months | Through study completion, an average of 1 year
  Survey questions asking about frequency, type (vaping vs. combustible); cannabis vs. tobacco; amount (relevant for vaping)

CONTACTS AND LOCATIONS:
Overall Officials: Karina M Shreffler, PhD, Principal Investigator — University of Oklahoma
Locations (1):
- OU Women's Health and Specialty Clinic, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Yes
Yes: There is a plan to make IPD and related data dictionaries available. All non-identifying IPD that underlie results in a publication will be made available to researchers upon request. Due to the small size of the sample, demographic characteristics will not be shared to eliminate the possibility of participant identification. Variables that will be shared include treatment group assignment, whether or not the pregnancy was unintended, maternal-fetal attachment scale, and self-reported smoking behavior.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Researchers will be able to request limited (e.g., non-identifying) IPD at the time of publication.
Access Criteria: Researchers must request IPD directly from PI Shreffler for access. Data published will be uploaded to FigShare, which allows the PI to securely provide a researcher with access to the data.

REFERENCES:
- [Background] Cranley MS. Development of a tool for the measurement of maternal attachment during pregnancy. Nurs Res. 1981 Sep-Oct;30(5):281-4. PMID 6912989
- [Background] Wise A, Geronimus AT, Smock PJ. The Best of Intentions: A Structural Analysis of the Association between Socioeconomic Disadvantage and Unintended Pregnancy in a Sample of Mothers from the National Longitudinal Survey of Youth (1979). Womens Health Issues. 2017 Jan-Feb;27(1):5-13. doi: 10.1016/j.whi.2016.10.006. Epub 2016 Nov 29. PMID 27913056
- [Background] Massey SH, Bublitz MH, Magee SR, Salisbury A, Niaura RS, Wakschlag LS, Stroud LR. Maternal-fetal attachment differentiates patterns of prenatal smoking and exposure. Addict Behav. 2015 Jun;45:51-6. doi: 10.1016/j.addbeh.2015.01.028. Epub 2015 Jan 20. PMID 25644587
- [Background] Shreffler KM, Tiemeyer S, Ciciolla L, Croff JM. Effect of a mindfulness-based pilot intervention on maternal-fetal bonding. Int J Womens Health. 2019 Jun 21;11:377-380. doi: 10.2147/IJWH.S203836. eCollection 2019. PMID 31417321